CLINICAL TRIAL: NCT02300272
Title: Modifiable Health Behaviors Associated With Time-of-Day Differences in Older Adults' Practice-Related Learning
Brief Title: Health Behaviors and Time-of-Day: Older Adult Cognitive Function
Acronym: OA-TIME
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400910
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Alteration of Cognitive Function; Ageing
Keywords: Practice-related learning; Sleep; Pain; Circadian Rhythm; Older Adults
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Typically healthy older adults: Adults 65 years and older with only common late-life medical conditions who will complete a screening that includes a Polysomnograph and assessment that includes Actiwatch.
  Interventions: Device: Polysomnograph; Device: Actiwatch

INTERVENTIONS:
Device: Polysomnograph — Participants will be screened for sleep disorders other than chronic insomnia with an in-home overnight sleep monitoring. Monitoring will consist of six electroencephalography (EEG) measures, two electrooculography (EOG), and chin electromyography (EMG) according to standard placements. Other channels will include oxygen saturation level, bilateral anterior tibialis EMG, heart rate (EKG), thoracic strain gauge, and a nasal/oral thermistor. A single night of polysomnography will be collected during the 2 weeks of assessment.
  Other Names: AURA Recording System, Grass Technologies
Device: Actiwatch — This device will be worn on the wrist for 14 continuous days to measure limb movements and ambient light.
  Other Names: Actiwatch-L, Mini Mitter

SUMMARY:
This is a single-center, observational study design. Enrolled participants will be typically, healthy older adults. Participants will complete daily computerized measures, in addition to continuously wearing an Actiwatch device. The study period will last 2 weeks. The objectives of the study are to examine the impact of sleep, pain, and circadian rhythm on practice-related learning in older adults at their preferred versus nonpreferred times of day.

DETAILED DESCRIPTION:
Participants will be asked to review the informed consent and consent to the study prior to any study procedure.

There are four stages to this study: 1. a telephone interview, 2. an in-person interview and completion of questionnaires, 3. an in-home single night sleep recording, and 4. two weeks of computerized cognitive testing, subjective sleep and pain recordings, and wearing a Actiwatch.

During the telephone interview, participants will be asked question about their age, sleep, pain, and medical/mental health history. At a second visit, participants will complete a more in-depth interview of their physical health, mental health, sleep, and pain history. They will complete a brief test of their cognitive functioning. They will also complete 4 questionnaires about their time of day preference and mood. At the third visit, participants will visit the University of Florida to be connected to a machine which will monitor their sleep. Participants will return home to sleep while still connected to the machine and will return the machine to the University of Florida the next day. Participants will complete brief computerized daily questionnaires of sleep and pain and cognitive testing in the morning and evening, and and wear an actigraph (wristwatch-like device) that measures arm movements and ambient light for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age of 65 years and older
* Able to read and speak English
* Completion of Morningness-Eveningness Questionnaire

Exclusion Criteria:

* Significant medical or neurological disorder
* Major psychopathology
* Pain disorder other than fibromyalgia or osteoarthritis
* Sleep disorder other than insomnia
* Cognitive impairment
* Psychotropic or other medications known to alter sleep
* Unable to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Typically, healthy older adults
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cognition as assessed by computerized neuropsychological testing | Morning and evening completion for 14 days
  Cognitive domains include processing speed, immediate memory, delayed memory, and executive function

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Robinson, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No